CLINICAL TRIAL: NCT06634485
Title: Correlation Between Spirometry ,diaphragmatic Ultrasound and Skeletal Muscle Mass in Patients with Chronic Obstructive Pulmonary Disease : Case Control Study
Brief Title: Spirometry ,diaphragmatic Ultrasound and Skeletal Muscle Mass in Patients with Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Mohamed Shazly, Principal Investigator, Assiut University
Other Study IDs: Ultrasound in COPD
Record Dates: First submitted 2024-08-21; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-08

CONDITIONS: COPD; Ultrasound Therapy; Complications
Keywords: COPD; Diaphragmatic Ultrasound; Spirometry; Skeletal Muscle Mass
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ultrasonography; Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- control group: This group include healthy volunteers who aged ≥ 40 years .
  Interventions: Device: ultrasound, spirometry
- study group: This include stable COPD Patients who will be diagnosed by GOLD 2024 and last excerbation ≥ 6weeks .
  Interventions: Device: ultrasound, spirometry

INTERVENTIONS:
Device: ultrasound, spirometry — Ultrasound assessment of
  1. diaphragmatic excursion:-the probe will be angled medially ,cranially , and dorsally so that the ultrasound beam reaches the posterior third of the diaphragm, in B-mode.Then, then M-mode exploration line will be placed perpendicular to the diaphragmatic dome to obtain maximum excursion .
  2. (Tdi) will be measured using a high-frequency linear probe (10 MHz) placed on (ZA).The probe will be angled perpendicular to the lateral chest wall and placed between the midaxillary and anterior axillary lines at the eighth or ninth intercostal space.
  3. Quadricep|rectus femoris muscle assessment will be done by placing the transducer perpendicular to the long axis of the thigh.
     * Spirometry:-will be performed thrice by experienced technicians at our pulmonary function laboratory. Patients will be asked to take a maximal inspiration and then to forcefully expel air for as long and as quickly as possible.

SUMMARY:
* The primary objective is to evaluate the use of diaphragmatic function and skeletal muscle mass by ultrasound as a tool to establish the diagnosis of COPD and assess the severity of the disease.
* The secondary objective is to compare diaphragmatic function, Skeletal muscle mass, and spirometry results in patients with COPD.

DETAILED DESCRIPTION:
* Chronic obstructive pulmonary disease (COPD) is a common preventable and treatable disease as per the Global Initiative for Chronic Obstructive Lung Disease (GOLD) and is characterized by persistent respiratory symptoms and airflow limitation that is due to airway and/or alveolar abnormalities usually caused by significant exposure to noxious particles or gases. According to the GOLD report, COPD is projected to be the third leading cause of death by 2020, and currently, it is the fourth .
* COPD is characterized by worsening dyspnea during movement . COPD restricts various activities of daily living due to shortness of breath, leading to poor quality of life and increased mortality and morbidity .
* COPD impairs the function of diaphragm which is the primary muscle of inspiration. Diaphragm provides 75% of the increase in lung volume during quiet inspiration .
* Movement of diaphragm during breathing is called diaphragm mobility. Movement of diaphragm from end-expiration to full inspiration is known as diaphragm excursion.
* Diaphragmatic mobility is lower in patients with COPD than in healthy individuals . Hence it is necessary to assess diaphragm function in inpatients and outpatients diagnosed with COPD during emergencies.
* Skeletal muscle dysfunction is a frequent and clinically relevant systemic manifestation of COPD that predicts morbidity and mortality independently from the severity of lung function impairment as judged by forced expiratory volume in 1 s (FEV1).Even in non cachectic patients with COPD, quadriceps strength is typically reduced by up to 30% compared with healthy elderly participants. Quadriceps strength independently predicts increased health-care utilization and mortality in COPD. While CT and magnetic resonance imaging (MRI) of the quadriceps have been studied in COPD, ultrasound use to assess limb muscle size has recently emerged as a newer, comparable, and noninvasive modality .
* Ultrasonography is a cost-effective, radiation-free, widely available, and real-time investigation.Many studies have proposed the possible use of ultrasonography to measure the diaphragmatic excursion .
* Spirometry is a noninvasive, easy, and valid tool for COPD assessment. There are established criteria based on spirometry, according to which COPD can be classified as mild, moderate, severe, and very severe .

There is a limited data about the association between spirometry, diaphragmatic excursion and skeletal muscle mass in patients with chronic obstructive pulmonary disease and further studies are needed

ELIGIBILITY:
Inclusion Criteria:

* Group A (control group):

  * This group include healthy volunteers who aged ≥ 40 years .
* Group B (study group):

  * This include stable COPD Patients who will be diagnosed by GOLD 2024 and last excerbation ≥ 6weeks .

Exclusion Criteria:

* Group A (control group):

  * Patients with disorders that may affect diaphragmatic function as

    1. Musculoskeletal / neurological disorders
    2. diaphragmatic eventration \ hiatus hernia
    3. morbid obesity
    4. recent thoracic/abdominal surgeries
    5. pregnancy; pleurodesis \fibrothorax.
* Group B (study group):-

  * Patients need for non- invasive ventilation.
  * Patients with disorders that may affect diaphragmatic function as

    1. Musculoskeletal / neurological disorders
    2. diaphragmatic eventration \ hiatus hernia
    3. morbid obesity
    4. recent thoracic/abdominal surgeries
    5. pregnancy; pleurodesis \fibrothorax

Ages: 41 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups will be enrolled in the study; the first group will include healthy volunteers who aged ≥ 40 years& the second group will include stable COPD Patients of the same age group
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
to study the correlation between diaphragmatic excursion and FEV1 | Day 1
  In the COPD group,The aim is to assess the correlation between diaphragmatic excursion and FEV1

SECONDARY OUTCOMES:
correlation between diaphragmatic muscle function , skeletal muscle mass and duration of hospital stay | Day 1
  correlation between diaphragmatic excursion measured by thoracic ultrasound in cm , quadriceps muscle thickness measured by ultrasound in cm and duration of hospital stay (in days)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shimizu M, Tozuka M. [Successful management of gingival and oral leukoplakia with non-smoking and vitamin B 2 butyrate esther]. Shikai Tenbo. 1982 Jul;60(1):201-4. No abstract available. Japanese. PMID 6957010
- [Background] Demain AL, Masurekar PS. Lysine inhibition of in vivo homocitrate synthesis in Penicillium chrysogenum. J Gen Microbiol. 1974 May;82(1):143-51. doi: 10.1099/00221287-82-1-143. No abstract available. PMID 4853060
- [Background] Winsey HS, Jones PF. Acute abdominal pain in childhood: analysis of a year's admissions. Br Med J. 1967 Mar 18;1(5541):653-5. doi: 10.1136/bmj.1.5541.653. No abstract available. PMID 6019663
- [Background] Youinou P, Pennec Y, Le Goff P, Ferec C, Morrow WJ, Le Menn G. Antiperinuclear factor in Sjogren's syndrome in the presence or absence of rheumatoid arthritis. Clin Exp Rheumatol. 1984 Jan-Mar;2(1):5-9. PMID 6335861
- [Background] Hodgkin JE. Preoperative evaluation of pulmonary function. Am J Surg. 1979 Sep;138(3):355-60. doi: 10.1016/0002-9610(79)90263-0. PMID 474874
- [Background] Bross ID, Natarajan N. Cumulative genetic damage in children exposed to preconception and intrauterine radiation. Invest Radiol. 1980 Jan-Feb;15(1):52-64. doi: 10.1097/00004424-198001000-00009. PMID 7353944
- [Background] Weisskopf B. Learning disorders in children: behavioral and emotional aspects of child and family. South Med J. 1969 Jul;62(7):811-5. No abstract available. PMID 5790674
- [Background] El-Halaby H, Abdel-Hady H, Alsawah G, Abdelrahman A, El-Tahan H. Sonographic Evaluation of Diaphragmatic Excursion and Thickness in Healthy Infants and Children. J Ultrasound Med. 2016 Jan;35(1):167-75. doi: 10.7863/ultra.15.01082. Epub 2015 Dec 17. PMID 26679203
- [Background] Schroll K. [Surgical removal of the upper 3d molars]. ZWR. 1986 Jun;95(6):630, 633-4, 637-9. No abstract available. German. PMID 3463040
- [Background] Taylor MA, Briggs GS, Baker KC, Cummings NJ, Pratt KA, Freedman RB, Goodenough PW. Expression of the pro-regions of papain and papaya proteinase IV in Escherichia coli and their inhibition of mature cysteine proteinases. Biochem Soc Trans. 1995 Feb;23(1):80S. doi: 10.1042/bst023080s. No abstract available. PMID 7758800
- [Background] Taggart SC. The healthy city. J R Coll Physicians Lond. 1998 Nov-Dec;32(6):568-71. No abstract available. PMID 9881315
- [Background] Kanareikin KF, Kukuev LA. [Soviet neuropathology during World War II 1941-1945 ( on the 50th anniversary of the outbreak of World War II)]. Zh Nevropatol Psikhiatr Im S S Korsakova. 1991;91(6):99-102. No abstract available. Russian. PMID 1664601
- [Background] Lopez AD, Shibuya K, Rao C, Mathers CD, Hansell AL, Held LS, Schmid V, Buist S. Chronic obstructive pulmonary disease: current burden and future projections. Eur Respir J. 2006 Feb;27(2):397-412. doi: 10.1183/09031936.06.00025805. No abstract available. PMID 16452599